CLINICAL TRIAL: NCT00011128
Title: Phase III Evaluation of the Role of Temporary Cessation of Antiretroviral Treatment and Resistance Testing-Based Selection of Antiretroviral Drugs in the Virologic Response to Salvage Therapy for Heavily Treatment-Experienced HIV-Infected Individuals Failing Current Antiretroviral Therapy
Brief Title: Salvage Treatment, Resistance Testing, and Withdrawal of Anti-HIV Drugs for HIV Patients Failing Current Anti-HIV Treatment
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5086; AACTG A5086; Substudy AACTG A5100s; Substudy AACTG A5104s
Record Dates: First submitted 2001-02-10; First posted 2001-08-31 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2004-05

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Resistance, Microbial; Microbial Sensitivity Tests; Salvage Therapy; Anti-HIV Agents; Viral Load; Treatment Experienced
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Behavioral: Antiretroviral Treatment Interruption

SUMMARY:
The purpose of this study is to test another way to control the amount of HIV in the blood (viral load).

Studies show that stopping all anti-HIV drugs for a time before switching to new anti-HIV drugs may improve the response in some individuals who are failing treatment. Other studies suggest a benefit if drug-resistance tests are used in selecting a new anti-HIV drug treatment. This study tests the effect of stopping anti-HIV drugs for a time before switching to anti-HIV drugs selected using drug-resistance test results.

DETAILED DESCRIPTION:
Virologic failure occurs in a large proportion of individuals receiving treatment with combination antiretroviral therapy. Studies suggest that treatment interruption prior to initiation of a multiple-drug rescue regimen may improve virologic response in individuals who have failed several prior antiretroviral regimens. Other studies suggest there is a virologic benefit derived from using genotypic or phenotypic resistance testing in selecting salvage therapy regimens for patients failing antiretroviral therapy. This study tests the hypothesis that salvage regimens selected on the basis of HIV-1 resistance genotype, phenotype [AS PER AMENDMENT 02/19/02: virtual phenotype], and treatment history will be more effective if there is a period of treatment interruption before initiating that regimen.

Patients continue their antiretroviral therapy until randomization. Based on the results of the pre-entry genotype and phenotype [AS PER AMENDMENT 02/19/02: virtual phenotype] tests and treatment history, an individualized salvage therapy regimen (not provided by the study) is selected by the site investigator(s). Additionally, patients start or continue maintenance therapy (not provided by the study) for opportunistic infections (OIs). Patients are randomized to 1 of 2 treatment arms. In Arm A, patients have antiretroviral treatment interruption for a period of 16 weeks (Step 1), followed by initiation of the [AS PER AMENDMENT 02/19/02: best available] salvage therapy regimen (Step 2). [AS PER AMENDMENT 02/19/02: Patients in Arm A will be placed immediately on their individualized salvage regimen before the end of the 16-week period of treatment interruption if their CD4 count falls below a defined threshold, or if they develop a new OI]. In Arm B, patients switch immediately to the salvage therapy regimen. [AS PER AMENDMENT 02/15/01: Patients who become pregnant during Step 1 of Arm A must be advised to begin their selected, individualized salvage therapy regimen or a modified salvage regimen. Patients who become pregnant during Step 2 of Arm A or Arm B have therapy evaluated and undergo any changes required by their pregnancy.] Patients in both arms are monitored for plasma HIV-1 RNA levels, CD4+ and CD8+ cell counts, and HIV drug resistance genotypes and phenotypes for a duration of 64 weeks from randomization. Patients in Arm A are also monitored for immune reactivation by measurement of T-cell subsets and plasma cytokines during treatment interruption. Patients may participate in a virology substudy (A5100s) and an immunology substudy (A5104s). [AS PER AMENDMENT 02/19/02: Patients who volunteer to participate in the substudies must be registered to the main study at the same time they are registered to a substudy.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-infected.
* Are likely to have drug-resistant HIV from having taken all types of anti-HIV drugs (protease inhibitors [PIs], nucleoside reverse transcriptase inhibitors [NRTIs], and nonnucleoside reverse transcriptase inhibitors [NNRTIs]), and having failed treatment prior to the current treatment for reasons other than toxicity.
* Are currently receiving anti-HIV treatment with at least 3 drugs. Low doses of ritonavir (100 to 200 mg twice daily) taken with 1 other PI is counted as a single PI.
* Are currently failing treatment due to a high viral load (amount of HIV in the blood).
* Have had a new anti-HIV drug combination selected.
* Are at least 18 years old.
* This study has been changed to remove CD4 counts as an inclusion criterion. In the previous version of the protocol, patients were required to have a CD4 count of 150 cells/ml or more within 42 days prior to study entry.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have stopped treatment for more than 4 weeks in the past 6 months.
* Are pregnant or breast-feeding.
* Have cancer that requires systemic treatment or radiation.
* Have received the following medications affecting the immune system within 14 days before entry: erythropoietin; Granulocyte Colony Stimulating Factor (G-CSF), including Granulocyte Macrophage Colony Stimulating Factors (GM-CSF); interleukins; or therapeutic HIV vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance A Benson, MD, Study Chair — University of Colorado, Denver; John Mellors, MD, Study Chair — University of Pittsburgh; Diane Havlir, MD, Study Chair — University of California, San Francisco
Locations (30):
- United States (29):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California, San Diego, San Diego, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of Hawaii, Honolulu, Hawaii
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Cornell Clinical Trials Unit - Chelsea Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Community Health Network Inc, Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Montaner JS, Harrigan PR, Jahnke N, Raboud J, Castillo E, Hogg RS, Yip B, Harris M, Montessori V, O'Shaughnessy MV. Multiple drug rescue therapy for HIV-infected individuals with prior virologic failure to multiple regimens. AIDS. 2001 Jan 5;15(1):61-9. doi: 10.1097/00002030-200101050-00010. PMID 11192869
- [Background] Lorenzi P, Opravil M, Hirschel B, Chave JP, Furrer HJ, Sax H, Perneger TV, Perrin L, Kaiser L, Yerly S. Impact of drug resistance mutations on virologic response to salvage therapy. Swiss HIV Cohort Study. AIDS. 1999 Feb 4;13(2):F17-21. doi: 10.1097/00002030-199902040-00001. PMID 10202819
- [Background] Hance AJ, Lemiale V, Izopet J, Lecossier D, Joly V, Massip P, Mammano F, Descamps D, Brun-Vezinet F, Clavel F. Changes in human immunodeficiency virus type 1 populations after treatment interruption in patients failing antiretroviral therapy. J Virol. 2001 Jul;75(14):6410-7. doi: 10.1128/JVI.75.14.6410-6417.2001. PMID 11413308
- [Background] Clevenbergh P, Durant J, Halfon P, del Giudice P, Mondain V, Montagne N, Schapiro JM, Boucher CA, Dellamonica P. Persisting long-term benefit of genotype-guided treatment for HIV-infected patients failing HAART. The Viradapt Study: week 48 follow-up. Antivir Ther. 2000 Mar;5(1):65-70. PMID 10846595
- [Background] Delaugerre C, Valantin MA, Mouroux M, Bonmarchand M, Carcelain G, Duvivier C, Tubiana R, Simon A, Bricaire F, Agut H, Autran B, Katlama C, Calvez V. Re-occurrence of HIV-1 drug mutations after treatment re-initiation following interruption in patients with multiple treatment failure. AIDS. 2001 Nov 9;15(16):2189-91. doi: 10.1097/00002030-200111090-00016. PMID 11684940
- [Result] Benson CA, Vaida F, Havlir DV, Downey GF, Lederman MM, Gulick RM, Glesby MJ, Wantman M, Bixby CJ, Rinehart AR, Snyder S, Wang R, Patel S, Mellors JW; ACTG A5086 Study Team. A randomized trial of treatment interruption before optimized antiretroviral therapy for persons with drug-resistant HIV: 48-week virologic results of ACTG A5086. J Infect Dis. 2006 Nov 1;194(9):1309-18. doi: 10.1086/508289. Epub 2006 Sep 22. PMID 17041858
- [Derived] Wang R, Bosch RJ, Benson CA, Lederman MM. Drug-resistant virus has reduced ability to induce immune activation. J Acquir Immune Defic Syndr. 2012 Dec 1;61(4):e60-3. doi: 10.1097/QAI.0b013e31827171d7. No abstract available. PMID 23138731